CLINICAL TRIAL: NCT00329823
Title: A Phase 2 Study of the Safety and Efficacy of Etanercept for the Therapy of Hydradenitis Suppurativa
Brief Title: Etanercept in Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-004555-19
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2006-05-25 (Estimated); Status verified 2006-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa, etanercept
MeSH Terms: conditions — Hidradenitis Suppurativa

INTERVENTIONS:
Drug: Etanercept sc 50mg per week for 12 weeks

SUMMARY:
The rationale of the protocol is based on the reported beneficiary results of case-patients by the administration of other anti-TNF drug (infliximab) in separate cases on the grounds of a probable autoimmune predisposition of the disease. The objective of this study is to clarify the potency of etanercept for the therapy of hidradenitis suppurativa.

DETAILED DESCRIPTION:
Hidradenitis suppurativa is a disorder of unknown etiology. Various hypotheses have implicated obesity, diabetes mellitus, genetic predisposition and tight clothing as probable contributing factors. Although patients are presenting with suppuration of their lesions, typical furuncles are absent (1). Administration of antibiotics offers transient relief of symptoms whereas therapies like androgens, isotretinoin and methotrexate have failed to disclose clinical benefit (2).

More than thirty out-patients with hidradenitis suppurativa are followed up at the clinic of the "Immunology of Infectious Diseases" of the ATTIKON University Hospital of Athens. None of them is presenting with diabetes mellitus and their CD4 cell counts are within normal limits. However, their testing for the function of monocytes is often abnormal. This test involves the isolation of monocytes and the ex vivo release of pro-inflammatory cytokines both without and after stimulation by bacterial endotoxins and lipoteichoic acid. Results have shown an increased baseline secretion and poor response of monocytes after stimulation.

Case reports with limited number of patients have disclosed clinical benefit of an other anti-TNF drug (infliximab) after one or two doses administration in hidradenitis suppurativa. These reports involve retrospective results of five patients (3) or single cases (4,5). The rationale of the administration of etanercept in hidradenitis suppurativa is based on the following data: a) etanercept has been proven effective for the management of psoriasis that is considered a skin disorder with autoimmune background (6); and b) laboratory findings of our patients with hidradenitis suppurativa point towards an altered immune response of their adaptive immunity (7).

Tumor necrosis factor (TNF) is a dominant cytokine in the inflammatory process of rheumatoid arthritis. Elevated levels of TNF are also found in the synovium of patients with psoriatic arthritis. Etanercept is a competitive inhibitor of TNF-binding to its cell surface receptors and thereby inhibits the biological activity of TNF. TNF and lymphotoxin are pro-inflammatory cytokines that bind to two distinct cell surface receptors: the 55-kilodalton (p55) and 75-kilodalton (p75) tumor necrosis factor receptors (TNFRs). Both TNFRs exist naturally in membrane-bound and soluble forms. Soluble TNFRs are thought to regulate TNF biological activity.

TNF and lymphotoxin exist predominantly as homotrimers, with their biological activity dependent on cross-linking of cell surface TNFRs. Dimeric soluble receptors such as etanercept possess a higher affinity for TNF than monomeric receptors and are considerably more potent competitive inhibitors of TNF binding to its cellular receptors. In addition, use of an immunoglobulin Fc region as a fusion element in the construction of a dimeric receptor imparts a longer serum half-life.

OBJECTIVE

The objective of this study is to clarify the potency of etanercept for the therapy of hidradenitis suppurativa.

RATIONALE

The rationale of the protocol is based on the reported beneficiary results of case-patients by the administration of other anti-TNF drug (infliximab) in separate cases on the grounds of a probable autoimmune predisposition of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of hidradenitis suppurativa
* Age > 16 years
* No presence of infections other then hidradenitis suppurativa.
* Disease activity index > 20
* Signed informed consent

Exclusion Criteria:

* Received any live (attenuated) vaccines within 4 weeks of enrolment visits
* Has a history of anti-cardiolipin antibodies associated with a thrombotic event
* Has a history of confirmed blood dyscrasias
* Has a significant active infection or any underlying diseases that could predispose subjects to infections (ie. Advanced or poorly controlled diabetes).
* Demonstrates liver function abnormality [SCOT, SGPT>2 X upper limit of normal]
* Has significant concurrent medical diseases including cancer or a history of cancer (other than resected cutaneous basal and squamous cell carcinoma) within 5 years of entering the enrollement period incompensated congestive heart failure, myocardial infarction within 12 months, unstable angina pectoris, uncontrolled hypertension, severe pulmonary disease, history of HIV infection, or central nervous system demyelinating events suggestive of multiple sclerosis.
* Has a history of known liver cirrhosis, fibrosis or fatty liver
* Has a history of any viral hepatitis
* Has renal disease (creatinine level > 175μmol/L)
* Has leucopenia (WBC <3500 x 106 /L)
* Has Thrombocytopenia (PLT's < 125 x 109 /L)
* Is pregnant or breast feeding.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Endpoints :
The disease activity index based on a calculated score.
The sum of the [diameter X severity] for each affected area.
Patient's global assessment of disease activity scores based on a VAS scale
of 1-10.
The number of newly presented lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Director — 4th Department of Internal Medicine, University of Athens, Greece; Helen Giamarellou, MD, PhD, Study Chair — 4th Department of Internal Medicine, University of Athens, Greece
Locations (1):
- 4th Department of Internal Medicine, University of Athens, Medical School, Athens, Greece

REFERENCES:
- [Background] Cusack C, Buckley C. Etanercept: effective in the management of hidradenitis suppurativa. Br J Dermatol. 2006 Apr;154(4):726-9. doi: 10.1111/j.1365-2133.2005.07067.x. PMID 16536817